CLINICAL TRIAL: NCT02309008
Title: A Randomized, Double-blind, Placebo-controlled Multiple Dosing Phase I Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics of PAC-14028 Cream After Transdermal Administration in Healthy Volunteers
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of PAC-14028 Cream in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: AP-TRPV1-PI-03
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics
MeSH Terms: interventions — N-(1-(3,5-difluoro-4-methanesulfonylaminophenyl)ethyl)-3-(2-propyl-6-trifluoromethylpyridine-3-yl)acrylamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): vehicle cream, dermal administration, multiple dosing
  Interventions: Other: Vehicle
- drug (Experimental): PAC-14028 cream, dermal administration, multiple dosing, dose escalation
  Interventions: Drug: PAC-14028

INTERVENTIONS:
Drug: PAC-14028 — Participants will receive PAC-14028 cream applied topically once a day for 9 days
  Other Names: PAC-14028 cream 0.1%; PAC-14028 cream 0.3%; PAC-14028 cream 1.0%
  Arms: drug
Other: Vehicle — Participants will receive vehicle cream applied topically once a day for 9 days
  Other Names: Vehicle cream
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate the safety/tolerability and pharmacokinetics of PAC-14028 cream after transdermal administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men aged 19 to 65 years at the time of screening
2. Whose weight is 50 kg or more, but less than 90 kg, and whose body mass index (BMI) is 18.0 kg/m^2 or more but less than 27 kg/m^2

   * BMI (kg/m^2) = weight(kg) /{height(m)}^2
3. Who doesn't have skin disease, skin damage (including tatoos or scars), or excessive hair in application area which can affect drug absorption
4. Who voluntarily decides study participation after receiving detailed explanation about the study and fully understanding it and who provides written consent for compliance with study requirement including proper contraception

Exclusion Criteria:

1. Who has clinically significant medical history or diseases involving liver, kidney, neurological system, respiratory system, endocrine system, urinary system, cardiovascular system,skin, psychical disorders or blood tumor
2. Who has a history of hypersensitivity or allergies to any drug (aspirin, antibiotics, etc)
3. Who has taken any prescribed drugs, herbal agents or crude drugs within 2 weeks before study drug administration, or who has taken any over-the-counter (OTC) drugs or vitamins within 1 week before the study drug initiation (Investigators will determine his eligibility by considering the effect of the drug on his safety or pharmacokinetic results in case other inclusion/exclusion criteria is satisfied.)
4. Who has drug abuse history or positive result at urine screening tests (cannabinoid, opioid, amphetamine, cocaine, barbiturate, benzodiazepine)
5. Who has smoked within 3 months before study drug administration (Smoker who has stopped smoking for more than 3 months before study drug administration is eligible to participate)
6. Who has confirmed positive at serological tests (HBs antigen, HCV antibody and HIV antibody)
7. Who consistently consumes alcohol
8. Who has participated in other clinical study within 8 weeks before study drug administration (however, the last dosing day is considered as the end of clinical study.)
9. Who has had bleeding or blood collection and donation over 400 mL within 8 weeks before study drug administration
10. Who donated whole blood within 2 months before study drug administration, who donated via plasmapheresis/plateletpheresis within 1 month before study drug administration, or who received a blood transfusion within 1 month before study drug administration
11. Whose vital sign measured at sitting position after resting at least 3 minutes is as following

    * Low blood pressure (Systolic pressure: less than 90 mmHg, Diastolic pressure: less than 60 mmHg)
    * High blood pressure (Systolic pressure: higher than 150 mmHg, Diastolic pressure: higher than 100 mmHg)
12. Who is determined ineligible for study participation by investigators for any reason including clinical lab test and ECG results.

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability (adverse events, abnormal vital signs, ECG test, clinical lab tests, Numerical pain recording scale) | Day 1~9, at specified time for each tests
  AE incidence pattern, abnormal findings in vital sign, ECG test, and clinical lab tests, Numerical pain recording scale

SECONDARY OUTCOMES:
Pharmacokinetics (Concentration of PAC-14028 in Blood; Cmax, AUC) | Day 1: 0 ~ 16h ; Day 2~8: 0h ; Day 9: 0 ~ 96h
  Concentration of PAC-14028 in Blood; Cmax, AUC

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital Clinical Trials Center, Seoul, South Korea